CLINICAL TRIAL: NCT03704129
Title: Evaluation of a 2-hour Educational Programme in Diaphragm Ultrasonographic Assessment
Brief Title: Educational Programme in Diaphragm Ultrasonographic Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paolo Navalesi (Other)
Responsible Party: Sponsor-Investigator, Paolo Navalesi, Prof, University Magna Graecia
Organization: University Magna Graecia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: US Diaphragm Learning
Record Dates: First submitted 2018-07-16; First posted 2018-10-12 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Educational Problems; Respiratory Muscle; Diaphragm Disease
Keywords: Diaphragm Ultrasound; Educational Programme

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Tutor" group (Experimental): After a theoretical part through the administration of a video-tutorial, a 10-point questionnaire will be administered to evaluate the level of learning for each participant. Every single participant will pass the test if he/she correctly answer to >70% of the questions. Those passing the test, will be randomized to two groups.
  The interventional group will access the practical training, during which each participant will be followed by a tutor who will interactively explain, using a healthy volunteer, how to perform the ultrasound scan of the diaphragm. The ultrasound will be performed on a healthy volunteer first by the tutor and then by the participants. During the exercise, each individual learner will be supervised by the tutor himself.
  Interventions: Other: Tutor
- "No tutor" group (No Intervention): This control group will directly perform the ultrasound examination of the diaphragm. The expert tutor will only show the learners how to use the various functions of the ultrasound, the linear and convex probes both in two-dimensional and in M-mode.

INTERVENTIONS:
Other: Tutor — The participants will access the practical training, during which each participant will be followed by a tutor who will interactively explain, using a healthy volunteer, how to perform the ultrasound scan of the diaphragm. The ultrasound will be performed on a healthy volunteer first by the tutor and then by the participants. During the exercise, each individual learner will be supervised by the tutor himself.
  Arms: "Tutor" group

SUMMARY:
Diaphragm ultrasound non-invasively explores the diaphragm function and it can be useful in several clinical situations. Diaphragm ultrasound is able to evaluate the cranio-caudal displacement of the diaphragm and its thickening fraction at the end of inspiration, in relation to the end-expiratory value.

While several studies have been conducted in the evaluation of educational programmes for echocardiography, to date data lack regarding this aspect in diaphragm ultrasonographic assessment.

Based on the experience gained in some specialization schools in Anaesthesia and Intensive Care, the investigators hypothesize that the participation in a two-hour course, including a theoretical part and a practical training, allows to acquire the appropriate theoretical and practical skills necessary to correctly perform the measurement of the diaphragm excursion and thickening fraction, compared to the theoretical lesson only, followed by a brief explanation by an expert tutor, on the practical use of the ultrasound.

The investigators hypothesized that the association of the theoretical part and of the practical training is able to obtain:

1. Passing the theoretical test with at least 70% of the correct answers;
2. The correct identification of the areas where the probe is affixed;
3. The appropriate measure of Diaphragmatic thickening and displacement.

DETAILED DESCRIPTION:
1. INTRODUCTION Diaphragm ultrasound non-invasively explores the diaphragm function and it can be useful in several clinical situations. Diaphragm ultrasound is able to evaluate the cranio-caudal displacement of the diaphragm and its thickening fraction at the end of inspiration, in relation to the end-expiratory value. These parameters provide useful data in the evaluation and management of patients affected by diaphragm dysfunction; moreover, they are gaining an increasing role in the evaluation of patients undergoing mechanical ventilation.

   To assess the diaphragm activity, clinicians use two different sonographic windows:

   i. to evaluate diaphragmatic thickness in the zone of apposition of the diaphragm to the rib cage. Physicians can assess thickening fraction between the 8th and 10th intercostal space, on the anterior or midaxillary line, 0.5-2 cm below the costophfrenic angle. The zone of apposition is the area of the chest wall where the abdominal contents reach the lower rib cage. In this area, the diaphragm is observed as a structure made of three distinct layers: a non-echogenic central layer bordered by two echogenic layers, the peritoneum and the diaphragmatic pleurae. To obtain adequate images of diaphragmatic thickness in M mode and 2D mode, a linear high-frequency probe (≥10 MHz) is necessary. The diaphragmatic thickness can be measured during quiet spontaneous breathing and during a maximal inspiratory and expiratory effort. An index of diaphragmatic thickening, the thickening fraction (TF) can be calculated using the M mode (TF = thickness at endinspiration - thickness at end-expiration/thickness at end-expiration). Diaphragmatic thickening fraction can be used as an index of diaphragmatic efficiency as a pressure generator. In normal individuals, there is a wide range of tdi at functional residual capacity (FRC), ranging between 1.8 to 3 mm. As lung volume increases from the residual volume (RV) to total lung capacity (TLC) there is a mean tdi increase of 54 % (range 42-78 %). Furthermore, the diaphragm also thickens during a maximal inspiratory pressure (Pimax) maneuver at FRC. A thickening ratio of 2.6 can be measured, dividing the diaphragmatic thickness during Pimax at FRC by the diaphragmatic thickness while relaxing at FRC.

   ii. the physicians can also assess the diaphragmatic displacement (or excursion) trough a 3.5-5 mHz phased array probe. The probe is placed immediately below the right costal margin in the mid-clavicular line or in the right anterior axillary line, and it is directed medially, cephalad and dorsally, in order that the ultrasound beam perpendicularly reached the hemi-diaphragm in its posterior third portion. After obtaining the best approach in two-dimensional mode, the displacement was measured in M-mode displaying the motion of the hemi-diaphragm along the selected line. In healthy subjects during spontaneous breathing, the inspiratory diaphragm excursion is 1.34 ± 0.18 cm.

   In patients undergoing assist mechanical ventilation, the thickening fraction is an indicator of inspiratory effort. While several studies have been conducted in the evaluation of educational programmes for echocardiography, to date data regarding this aspect in diaphragm ultrasonographic assessment lack.
2. AIM OF THE STUDY

Based on the experience gained in some specialization schools in Anesthesia and Intensive Care, the investigators hypothesize that the participation in a two-hour course, including a theoretical part and a practical training, allows to acquire the appropriate theoretical and practical skills necessary to correctly perform the measurement of the diaphragm excursion and thickening fraction, compared to the theoretical lesson only, followed by a brief explanation by an expert tutor, on the practical use of the ultrasound. The investigators hypothesized that the association of the theoretical part and of the practical training is able to obtain:

1. Passing the theoretical test with at least 70% of the correct answers;
2. The correct identification of the areas where the probe is affixed;
3. The appropriate measure of diaphragmatic TF and displacement.

3. MATERIALS AND METHODS Participants will be randomized into two groups similar for age and gender. First of all, a theoretical part will be conducted through the administration of a video-tutorial to both groups, aimed to teach of ultrasonographic basic principles, of sonographic windows and of the anatomical reference points for the diaphragmatic ultrasonography. At the end of the video, a 10-point questionnaire will be administered to evaluate the level of learning for each participant.

Every single participant will pass the test if he/she correctly answers to at least the 70% of the questions. Those passing the test will be randomized to two groups. Participants will be randomly assigned to one of the two groups using opaque, sealed, numbered envelopes. The investigators will use a computer-generated randomization sequence, generated by an independent biostatistician who is not otherwise involved in the trial. The envelopes will be kept in head of nurses offices in every institution's critical care unit. The researcher will distribute the envelopes to participants, which will independently open it. Participants will communicate the random group allocation to the researcher who will assign the participant to the study group.

The first group will access the practical training, during which each participant will be followed by a tutor who will interactively explain, using a healthy volunteer, how to perform the ultrasound scan of the diaphragm. The ultrasound will be performed on a healthy volunteer first by the tutor and then by the participants. During the exercise, the tutor himself will supervise each individual learner.

The second group will directly perform the ultrasound examination of the diaphragm. The expert tutor will only show the learners how to use the various functions of the ultrasound, the linear and convex probes both in two-dimensional and in M-mode.

The tutors assigned to both groups will have proven experience in thoracic ultrasound. In order to standardize the practical teaching of the technique, the tutors will meet telematically by agreeing the modalities of the training and / or administration of the basics on the use of the ultrasound.

To evaluate the learning, each participant of both groups will perform the ultrasound scan of the diaphragm in both acoustic windows and acquire the images on the healthy volunteer. The tutor will verify the correctness of the acquired images and make the measurements.

A classroom helper will record the measurements taken and make the scanned image available again for a new measurement. Therefore, on the same image, the participant, who will not know the measurements performed by the tutor, will perform his own measurement, the results of which will be recorded by the person in charge of the classroom. This procedure will be carried out both for the measurement of the excursion and for that of the thickening fraction.

If the participant fails to correctly display the diaphragm in one of the two windows, the result will be negative. Those who will identify the diaphragm in both windows will be admitted to the next step and will be able to measure the diaphragmatic displacement and the diaphragmatic thickening fraction. The result will be considered positive if the learner will obtain measurement values for thickening fraction that deviate from those performed by the expert tutor at most 20% and diaphragmatic displacement values that deviate from the values obtained by the tutor to a maximum of +/- 2 mm.

A. Study design Multicenter randomized controlled study.

B. Population 58 students for each of the two groups, for a total of 116 volunteers, enrolled between medical and surgical students, health professions, specializing in medical-surgical disciplines who have no experience in the field of ultrasound and are divided into two groups, of which one will receive both the theoretical lesson and the practical training, while the other at the end of the theoretical lesson will receive only general notions about the practical use of the ultrasound.

C. Statistical analysis Based on the above considerations, at the end of the course, a difference is expected between groups receiving the practical training compared and control, in terms of achievement of the outcome equal to at least 30%.

ELIGIBILITY:
Inclusion Criteria:

* 116 students with no experience in the field of ultrasound

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic skills - Thickening Fraction | Soon after the video-tutorial (within 30 minutes), when participants perform diaphragm ultrasound
  Measurement of thickening fraction. If measurements will deviate from those recorded by the expert within the 20% of the value, the result will be considered positive
Ultrasonographic skills - Diaphragm Displacement | Soon after the video-tutorial (within 30 minutes), when participants perform diaphragm ultrasound
  Measurement of Diaphragm Displacement. If students' measurements will deviate from those recorded by the expert within the +/- 2 mm, the result will be considered positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Eugenio Garofalo, Catanzaro, CZ, Italy

IPD SHARING:
Plan to Share IPD: Yes
All individual, de-identified participant data will be shared after motivated request by e-mailing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the anticipated end of the trial
Access Criteria: Motivated request by e-mailing

REFERENCES:
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Umbrello M, Formenti P, Longhi D, Galimberti A, Piva I, Pezzi A, Mistraletti G, Marini JJ, Iapichino G. Diaphragm ultrasound as indicator of respiratory effort in critically ill patients undergoing assisted mechanical ventilation: a pilot clinical study. Crit Care. 2015 Apr 13;19(1):161. doi: 10.1186/s13054-015-0894-9. PMID 25886857
- [Derived] Garofalo E, Bruni A, Pelaia C, Landoni G, Zangrillo A, Antonelli M, Conti G, Biasucci DG, Mercurio G, Cortegiani A, Giarratano A, Vetrugno L, Bove T, Forfori F, Corradi F, Vaschetto R, Cammarota G, Astuto M, Murabito P, Bellini V, Zambon M, Longhini F, Navalesi P, Bignami E. Comparisons of two diaphragm ultrasound-teaching programs: a multicenter randomized controlled educational study. Ultrasound J. 2019 Oct 3;11(1):21. doi: 10.1186/s13089-019-0137-4. PMID 31578700